CLINICAL TRIAL: NCT04583982
Title: ImmuneSense™ COVID-19 Study
Status: Completed | Type: Observational
Sponsor: Adaptive Biotechnologies (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00781
Record Dates: First submitted 2020-10-07; First posted 2020-10-12 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Disease (COVID-19); SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Study Arm SARS-CoV-2 negative and positive samples
  Interventions: Other: T-Detect™ SARS-CoV-2 Assay

INTERVENTIONS:
Other: T-Detect™ SARS-CoV-2 Assay — T-Detect™ SARS-CoV-2 Assay is an investigational device that is indicated to assess T-cell immune response to SARS-CoV-2 via the testing of blood samples from patients with signs and symptoms of suspected COVID-19. These results will not be shared with the participant.

SUMMARY:
Coronavirus disease is of an urgent global priority. The purpose of ImmuneSense™ COVID-19 study is to evaluate the clinical performance and to provide data for clinical validation for the T-Detect™ SARS-CoV-2 (previously referred to as immunoSEQ Dx SARS-CoV-2) Assay in support of Adaptive's Emergency Use Authorization (EUA) request for T-Detect™ SARS-CoV-2 and secondary aims. This assay is intended to detect immune response to the virus that causes coronavirus disease (COVID-19), SARS-CoV-2. This is critically important because the immune system may be able to tell us important information about how our own bodies detect and respond to the disease that current tests cannot.

DETAILED DESCRIPTION:
Comprehensive diagnostic testing has an important role to play in the control and containment of the current pandemic. Adaptive Biotechnologies Corporation (Adaptive) has developed an immunosequencing technology, called immunoSEQ®, which utilizes polymerase chain reaction (PCR) and next-generation sequencing (NGS) to identify and quantify rearranged T-cell receptor (TCR) gene sequences from peripheral blood, collectively referred to as the T-cell repertoire. The T-cell repertoire can be further analyzed using indication-specific algorithms that are based on disease-associated TCR sequences.

Adaptive has developed a clinical test called T-Detect™ SARS-CoV-2, which is intended to identify a T-cell response to the SARS-CoV-2 virus, indicating recent or prior infection. In this investigational study, Adaptive plans to clinically validate samples acquired from patients with COVID-19 and present results for an eventual EUA-submission for the T-Detect™ SARS-CoV-2 Assay. T-Detect™ SARS-CoV-2 is a single-site assay performed at Adaptive Biotechnologies Corporation.

ELIGIBILITY:
Inclusion Criteria

Participants must satisfy the following criteria to be enrolled in the study:

* Currently symptomatic individuals who are being tested for SARS-CoV-2 infection by nasopharyngeal swab
* Male and female participants of any race and ethnicity between 18 to 89 years of age (inclusive) at the time of enrolling in the study
* Must be able to communicate with the investigator, understand, and comply with the requirements of the study

Exclusion criteria

The presence of any of the following will exclude a participant from enrollment:

* Asymptomatic individuals who are being tested for SARS-CoV-2 infection
* Prior confirmed diagnosis of COVID-19
* Any person who cohabitated with another individual with known COVID-19
* Protected populations including minors, pregnant women, prisoners, mentally disabled persons, and wards-of-the state
* Any significant condition, laboratory abnormality, or psychiatric illness that would prevent the participant from safely participating in the study
* Donated more than 500cc or 1 pint of blood in the past 60 days prior to the blood draw
* Participation in a COVID-19/SARS-CoV-2 study or received a COVID-19 vaccine, antibody, or other COVID-19 therapeutic Investigational drug or compound that will impact results of the study at the discretion of the investigator, such as but not limited to a COVID-19 antibody, therapeutic, or other medication that will impact the person's immune system

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants include male and female participants, of any race and ethnicity, ages 18-89.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Demonstrate clinical agreement of T-Detect™ SARS-CoV-2 Assay | Initial Visit
  To demonstrate the clinical agreement of the T-Detect™ SARS-CoV-2 Assay in participants with a positive and negative result from an EUA approved RT-PCR assay.

CONTACTS AND LOCATIONS:
Overall Officials: Namita Singh, MD, Study Director — Medical Director, Clinical Development
Locations (1):
- Adaptive Biotechnologies Clinical Investigational Site, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No